CLINICAL TRIAL: NCT05299580
Title: "Dabrafenib and Trametinib in Circulating Free DNA BRAFV600 Mutated Metastatic Melanoma Patients: a Prospective Phase II, Open Label, Multicentre Study - (Bioliquid TAILOR Study - BIOTAILOR)"
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Fondazione Melanoma Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-TAILOR
Record Dates: First submitted 2022-02-23; First posted 2022-03-29 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Patients will be treated with Dabrafenib 150 mg bid and Trametinib 2mg qd. Each cycle is 28 days and the treatment will be continued until documented disease progression, unacceptable toxicity, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons.
  Interventions: Drug: dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: dabrafenib — Dabrafenib 150 mg bid
Drug: Trametinib — Trametinib 2mg qd

SUMMARY:
There is evidence from cohort studies and metanalysis that a shift from BRAFWT to BRAF mutated melanomas can occur (Colombino JCO 2012, Valchis EJC 2017). Based on previous studies we expect that 15% of tissue BRAF WT patients treated with anti PD-1 will become circulating free DNA BRAF (CfDNA BRAF) mutation-positive and, at progression, they will be elegible to be treated with dabrafenib/trametinib. We aimed to design a clinical phase II trial in order to evaluate the activity of Dabrafenib and Trametinib in patients with Tissue BRAFWT signature and a molecular shift to circulating free DNA BRAF mutated positive melanomas upon progression to anti PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥ 18 years;
2. Histologically confirmed stage III (unresectable) or stage IV melanoma;
3. Tissue BRAFWT signature and a molecular shift to circulating free DNA BRAF mutated positive melanomas upon progression to anti PD-1 therapy;
4. Tumor biopsy, if feasible, to confirm the BRAFV600 mutation at progression;
5. Previous adjuvant treatment, including checkpoint inhibitors anti CTLA-4, anti PD- 1/PDL-1 is allowed, except for stage IV (if completed at least 6 months prior to enrollment, and all related adverse events have either returned to baseline or stabilized). BRAF inhibitor treatment in adjuvant setting is not permitted;
6. Last previous treatment for metastatic disease MUST BE Anti-PD1 as single agent;
7. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels;
8. Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria;
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2 (see Appendix II);
10. Female subjects of childbearing potential must have a negative pregnancy test result at baseline and must practice two highly effective methods of contraception for the duration of the study, EOT, at 30-day and 150-day safety follow up;
11. Sexually active males must agree to use effective contraception methods throughout treatment and for 150 days after stopping treatment and should not father a child in this period. A condom is required to be used by vasectomized men as well during intercourse in order to prevent delivery of the drug via semen;
12. Adequate baseline organ function
13. Life expectancy of at least 3 months;
14. Ability to understand study-related patient information and provision of written informed consent for participation in the study.

Exclusion Criteria:

1. Symptomatic brain metastases;
2. History of another malignancy, exception: subjects who have been disease-free for 3 years, (i.e. subjects with second malignancies that are indolent or definitively treated at least 3 years ago) or subjects with a history of completely resected nonmelanoma skin cancer;
3. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy including:

   * Presence of predisposing factors to RVO or central serous retinopathy (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or
   * Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or central serous retinopathy such as: i. Evidence of new optic disc cupping; ii. Evidence of new visual field defects on automated perimetry; iii. Intraocular pressure >21 mmHg as measured by tonometry.
4. A history of clinically significant or active interstitial lung disease or pneumonitis;
5. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures;
6. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted);
7. A history or evidence of cardiovascular risk including any of the following:

   * Current LVEF < LLN;
   * A QT interval corrected for heart rate using the Bazett's formula >480 msec;
   * A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with atrial fibrillation controlled for > 30 days prior to enrollment are eligible;
   * A history (within 6 months prior to enrollment) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty;
   * A history or evidence of current >= Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines;
   * Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy;
   * Patients with intra-cardiac defibrillators or permanent pacemakers;
   * Known cardiac metastases;
   * Abnormal cardiac valve morphology (> grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study;
   * Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia), long QT syndrome or taking medicinal products known to prolong the QT interval.
8. Female subjects who are pregnant (positive pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control;
9. Inability to regularly access site facilities for logistical or other reasons;
10. History of poor co-operation, non-compliance with medical treatment, or unreliability;
11. Participation in any interventional drug or medical device study within 30 days prior to treatment start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | From day 1 up to 24 months Every 12 weeks
  proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From day 1 up to 24 months Every 12 weeks
  the time from the date of first administration of therapy and the date of evidence of progression or death
Overall Survival | from 28 days from baseline up to 24 months
  the time from the date of first administration of therapy and the date of death from any cause.
Safety - NCI CTC-AE (Version 5.0) | up to 24 months
  Will be used to evaluate the clinical safety of the treatment in this study; patients will be assessed for AEs at each clinical visit and as necessary throughout the study.
QoL | From day 1 up to 24 months Every 12 weeks
  the 30-item European Organisation for Research and Treatment of Care quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - IRCCS - Istituto Scientifico Romagnolo per la Cura e lo Studio dei Tumori (I.R.S.T) S.r.l., Meldola, Forlì-Cesena
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - National Institute of Cancer, Bari
  - Università degli Studi di Bari Aldo Moro, Bari
  - AOU Sant'Orsola-Malpighi, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - Azienda Sanitaria Ospedaliera S. Croce e Carle, Cuneo
  - IRCCS San Martino - IST, Genova
  - Fondazione I.R.C.C.S. Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria di Modena, Modena
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Giovanni Pascale", Naples
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Universitaria - Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata di Udine, Udine